CLINICAL TRIAL: NCT01973946
Title: Telephone Linked Care: An IT Enabled Integrated System for Cancer Symptom Relief
Brief Title: Cancer Symptom Monitoring Telephone System With Nurse Practitioner (NP) Follow up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kathleen Mooney, Principal Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17472; 5R01CA120558 (NIH)
Record Dates: First submitted 2013-10-22; First posted 2013-11-01 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Cancer
Keywords: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (No Intervention): Patients in the usual care group called the automated monitoring system daily to report presence, severity, and distress for 11 common symptoms. The attentional control group received equivalent contact time with the automated system including identical voice and assessment questions. Patients did not hear self-care messages during the call and the data were not available for clinical action by the study nurse practitioner. Patients were told on every phone call to call their oncology providers if they had concerns about their symptoms which is usual care for symptom follow up in oncology.
- Symptom Alert and Coaching (Experimental): Patients in the Symptom Alert and Coaching arm called the automated monitoring system daily to report presence, severity, and distress on 11 symptoms. The system provided automated self care coaching based on the symptoms reported and automatically generated alerts to the study NP if symptoms exceeded preset thresholds. Two thresholds were set: a simple alert when severity or distress was 4 or greater on a 10 point scale and trend alerts based on a pattern of moderate severity over several days.
  The alerts went into a case management site. The study NP logged into the system daily and responded to the alerts within 24 hours by calling patients to further assess the symptoms and to intensify symptom treatment using evidence based guidelines.
  Interventions: Other: Symptom Alert and Coaching

INTERVENTIONS:
Other: Symptom Alert and Coaching — Patients heard self-care messages when they reported a symptom was present. The Symptom Alert and Coaching intervention alerted study nurse practitioners of unresolved symptoms daily. The NPs responded to all alerts generated by patients and using evidence based guidelines, called patients to further assess and to intensify symptom treatment.
  Arms: Symptom Alert and Coaching

SUMMARY:
The purpose of this prospective trial is to test a daily telephone based automated symptom monitoring and response system to track and further treat unrelieved symptoms for patients living at home during chemotherapy treatment as compared with usual care which consists of patients calling their oncology provider for symptom concerns.

DETAILED DESCRIPTION:
The purpose of this prospective trial is to test a daily telephone based automated symptom monitoring and response system to track and further treat unrelieved symptoms for patients living at home during chemotherapy treatment as compared with usual care which consists of patients calling their oncology provider for symptom concerns. For the intervention group, the monitoring system is paired with automated delivery of self-care suggestions tailored to the specific symptom profile the patient reported and also automatically 'alerts' the study oncology nurse practitioner about unrelieved symptoms. The nurse practitioner, utilizing national evidence based symptom guidelines for symptoms at moderate to severe levels calls the patient and further assesses and intensifies symptom treatment. The usual care group called the system daily and reported similar data but did not receive self-care coaching or notification of unrelieved symptoms to the study nurse practitioner. On every call, the usual care group was told to follow the standard procedure of calling their oncology providers for symptom concerns. The specific aims of the study are to test whether the symptom monitoring intervention reduces presence, severity and distress of 11 symptoms. The symptoms monitored in the project were nausea/vomiting, pain, sore mouth, numbness & tingling, diarrhea, trouble thinking, trouble sleeping, changes in appearance, depressed mood, anxiety, and fatigue. Secondary outcomes tested whether the intervention improved functional performance and decreased interference with activity when compared with the usual care attentional control group. Other aims compare self care strategies utilized and their perceived effectiveness and document patient satisfaction with the monitoring system.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age 18 or over)
* Have a histological diagnosis of cancer
* a life expectancy of at least 3 months and cognitively able to participate
* Beginning a new course of chemotherapy that is planned for a minimum of 3 cycles;
* care is under the direction of one of the 8 designated provider teams;
* English speaking;
* has access to a telephone on a daily basis and is able to use the phone unassisted as verified by the study staff during participant orientation.

Exclusion Criteria:

* patients who are receiving concurrent radiation therapy (as they would have daily contact with the health care system);
* patients who see the provider team for recommendation of a chemotherapy regimen but treatment is then administered at a different site by other providers.
* Patients receiving therapy agents that result in a drug related fever or therapy agents that are not anticipated to cause any of the 11 symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2007-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Patient reported symptom levels | Daily patient reports of symptom levels were made for an entire new course of chemotherapy or 6 months whichever occurred first.
  During daily automated calls, patients provided information about common chemotherapy symptoms on a 0-10 scale.

SECONDARY OUTCOMES:
Medical Encounters Telephone Interview | Each week patients reported during the daily symptom monitoring call whether they had a medical encounter for an entire new course of chemotherapy or 6 months whichever occurred first.
  Each week patients reported during their daily phone calls whether or not they had been in contact with a health care provider, were seen in an emergency department or urgent care facility, or had an unscheduled hospitalization. If they reported they did have a medical encounter, the research staff would call and conduct a short telephone interview to collect data about the nature of the medical encounter including whether the medical encounter was related to the symptoms being monitored.
Patient reported symptom related interference with daily activities | Reported daily for an entire new course of chemotherapy or 6 months whichever occurred first.
  This is a one item question asked daily during the symptom monitoring call about the level of interference their symptoms had on their daily activities (0-10 scale).
SF-36 Functional Status | Monthly for an entire new course of chemotherapy or 6 months whichever occurred first.
  Functional status was measured monthly using the SF-36.
Work interference | Reported daily for an entire new course of chemotherapy or 6 months whichever occurred first.
  For patients who indicated they worked during their treatment, the system asked daily if they missed work if it was a regular workday.
Work Limitations Questionnaire | Monthly for an entire new course of chemotherapy or 6 months whichever occurred first.
  The 25 item patient-reported Work Limitations Questionnaire was used to measure work performance.

OTHER OUTCOMES:
Patient End of Study Telephone Interview | Administered once, at the end of the patients' participation in the study which was following an entire new course of chemotherapy or 6 months whichever occurred first.
  An End of Study Telephone Interview was conducted at the end of a patient's participation in the project to obtain data on patient satisfaction with the symptom monitoring system and to obtain suggestions for improvement of the system.
Evaluation of automated and other self care strategies used and their effectiveness | Weekly for an entire new course of chemotherapy or 6 months whichever occurred first.
  The symptom monitoring system tracked when an intervention participant heard a self care strategy during the course of the week. Each week patients would report on how helpful (1-10 scale) the automated self care measures were for the specific symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen H Mooney, PhD, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - University of Utah Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mooney K, Beck SL, Wilson C, Coombs L, Whisenant M, Moraitis AM, Sloss EA, Alekhina N, Lloyd J, Steinbach M, Nicholson B, Iacob E, Donaldson G. Assessing Patient Perspectives and the Health Equity of a Digital Cancer Symptom Remote Monitoring and Management System. JCO Clin Cancer Inform. 2024 Jul;8:e2300243. doi: 10.1200/CCI.23.00243. PMID 39042843
- [Derived] Moraitis AM, Iacob E, Wong B, Beck SL, Echeverria C, Donaldson G, Mooney K. Pairing automated exercise coaching with patient-reported symptom monitoring: A way to nudge exercise uptake during cancer treatment? Support Care Cancer. 2024 Apr 1;32(4):258. doi: 10.1007/s00520-024-08450-1. PMID 38558321
- [Derived] Mooney KH, Beck SL, Wong B, Dunson W, Wujcik D, Whisenant M, Donaldson G. Automated home monitoring and management of patient-reported symptoms during chemotherapy: results of the symptom care at home RCT. Cancer Med. 2017 Mar;6(3):537-546. doi: 10.1002/cam4.1002. Epub 2017 Jan 30. PMID 28135050